CLINICAL TRIAL: NCT00362817
Title: Phase I/II Multicenter Trial of Intra-Arterial Carboplatin and Oral Temozolomide for the Treatment of Recurrent and Symptomatic Residual Brain Metastases.
Brief Title: Carboplatin and Temozolomide (Temodar) for Recurrent and Symptomatic Residual Brain Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0428
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Brain Tumor; Brain Metastases
Keywords: Recurrent; Symptomatic
MeSH Terms: conditions — Brain Neoplasms; Recurrence | interventions — Carboplatin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide & Intra-Arterial (IA) carboplatin (Experimental): Patients will be administered Temozolomide orally once a day for 5 consecutive days and and will receive Intra Arterial Carboplatin
  Interventions: Drug: carboplatin; Drug: temozolomide

INTERVENTIONS:
Drug: carboplatin — IA carboplatin 200 mg/m2/day for each arterial injection on days 1 and 2.
  Other Names: Paraplatin; CBDCA
Drug: temozolomide — 150 mg/m2/day orally Days 1-5. Treatment cycles to be repeated every 4 weeks.
  Other Names: Temodar

SUMMARY:
Purpose: The primary objective of this study is to determine if chemotherapy with carboplatin and temozolomide significantly affects the response rates, or size of disease, in patients with brain metastases, originating from cancer in other parts of the body, compared to patients who have already been treated with radiation. Survival, causes of death, recurrence of disease in the central nervous system, toxicity, and quality of life will all be measured as secondary objective in this study.

DETAILED DESCRIPTION:
Rationale: Surgery and radiation are often used as treatments for brain metastases, or tumors in the brain that originate from other parts of the body. It is currently unknown whether patient survival or time to progression would experience additional benefits through the addition of chemotherapy. Previous research does appear to suggest that a chemotherapy regimen may improve outcomes of patients with brain metastases previously treated with radiation. The current study further evaluates this research question by providing patients with recurrent or symptomatic residual brain metastases with carboplatin and temozolomide, two chemotherapy agents. Temozolomide has demonstrated clinical antitumor efficacy against malignant gliomas and has been tested with some efficacy against several other types of cancer. This drug appears to have less adverse effects compared to other commonly used cancer drugs. Recent research indicates that temozolomide also has some efficacy against brain metastases. In addition, previous research indicates carboplatin's lack of severe toxicity in patients with this disease.

Treatment: Study participants will be treated with carboplatin and temozolomide. Carboplatin will be administered through intravenous infusions. Temozolomide will be given through oral pills. Before these drugs are administered, study participants will undergo a pre-treatment evaluation with physical and neuropsychological examinations, neuro-imaging, laboratory tests, quality of life assessment, and other procedures. Carboplatin will be given for two consecutive days. Temozolomide will be taken by study participants daily for five consecutive days. Both of these treatment schedules will be repeated every 28 days. Several tests and exams will be given throughout the study to closely monitor patients. Study treatments will be discontinued due to disease growth or unacceptable adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed systemic cancer

Exclusion Criteria:

* Pregnant
* Known CNS meningeal involvement with cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Newton, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients had received prior systemic chemotherapy for the primary tumor
Groups:
- Temozolomide & Intra-Arterial (IA) Carboplatin: Patients will be administered Temozolomide orally once a day for 5 consecutive days and and will receive Intra Arterial Carboplatin
  temozolomide : 150 mg/m2/day orally Days 1-5. Treatment cycles to be repeated every 4 weeks.
  carboplatin : IA carboplatin 200 mg/m2/day for each arterial injection on days 1 and 2.
Period: Overall Study
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 52 [34 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Affects of Response Rate of Chemotherapy With Intra-arterial Carboplatin and Oral Temozolomide
Description: Response was evaluated by MRI Criteria (MacDonald Criteria). The MacDonald criteria for determining tumor progression is determined through assessing the increase in size of an enhancing tumor on consecutive MRI scans and clinical assessment. Complete response occurs when there is a disappearance of all enhancing tumor on consecutive MRI scans at least one month apart. Partial response occurs at a >50% reduction in size of enhancing tumor on consecutive MRI scans at least one month apart. Progressive disease occurs when there is a >25% increase in size of enhancing tumor on consecutive MRI scans. Stable disease occurs in all remaining situations.
Time Frame: up to 1 year
Measure: Number; unit: percentage of patients with response
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 14
percentage of patients with response | 42.8

2. Secondary Outcome: Analyze Patients Time to Progression
Description: Responses to treatment was determined by comparing new enhanced MRI scans with those obtained at the previous evaluation (i.e., 2 treatment cycles ago) or with the pre-IA chemotherapy baseline scan, if it is the first follow-up MRI scan during treatment.
  MRI is the neuro-imaging modality of choice, since it is more accurate than CT for small tumors, multiple tumors, and tumors in the posterior fossa.58 The methodology used (techniques and equipment) must be identical for all scans. Lesions should be measured as the largest diameter seen on scan and the largest diameter perpendicular to that dimension.
Time Frame: up to 60 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 14
weeks | 22.6 [8 to 60]

3. Secondary Outcome: Determine the Overall Survival of Patients
Description: From the time of protocol initiation
Time Frame: up to 64 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 14
weeks | 25.2 [12 to 64]

4. Secondary Outcome: Determine the Cause of Death of Patients After Treatment
Description: To determine the cause of death (i.e., CNS tumor versus systemic disease progression) in patients after treatment.
Time Frame: up to 1 year
Measure: Number; unit: patients
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 14
patients
  CNS tumor | 0
  Systemic disease progression | 7

5. Secondary Outcome: The Incidence and Severity of Centeral Nervous System (CNS) Toxicities
Description: To determine the incidence and severity of CNS toxicity in patients treated with intra-arterial carboplatin and oral temozolomide.
Time Frame: up to 24 weeks
Measure: Number; unit: patients
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 14
patients | 0

6. Secondary Outcome: Quality of Life Assessment
Description: To determine the impact of treatment on quality of life.
Time Frame: up to 2 years
Population: Quality of Life Assessment was not done.
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Temozolomide & Intra-Arterial (IA) Carboplatin
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes